CLINICAL TRIAL: NCT04372511
Title: Evaluation of Pain and Patient Satisfaction Using Binaural Beats in Patients Submitted to Colonoscopy
Brief Title: Use of Binaural Beats for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Responsible Party: Principal Investigator, Alessandro Tani, Principal Investigator, Azienda USL Toscana Nord Ovest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: usl toscana nordovest
Record Dates: First submitted 2020-04-26; First posted 2020-05-04 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Pain
Keywords: Binaural Beats; Colonscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binaural Beats (Experimental): Group A : use of stereo headphones that generate sound with Binaural Beats at acoustic frequencies of 256 Hz in one ear and 260 Hz in the opposite ear producing a binaural beat of 4 Hz with a white background noise
  Interventions: Device: Binaural Beats
- No sounds (No Intervention): Group B : use of stereo headphones with a white background noise

INTERVENTIONS:
Device: Binaural Beats — Device: Sound with Binaural Beats at acoustic frequencies of 256 Hz in one ear and 260 Hz in the opposite ear producing a binaural beat of 4 Hz with a white background noise
  Arms: Binaural Beats

SUMMARY:
Investigators verify the effectiveness of "binaural beats" to reduce pain during colonoscopy .

DETAILED DESCRIPTION:
Colonoscopy is a disturbing and painful procedure, so whenever possible it is performed in sedation. Although the use of sedative drugs is effective in relieving anxiety and pain such drugs can cause significant side-effects.

This study examines the effect of Binaural Beats stimulation on pain perception during colonscopy.

Binaural Beats is a simple technique, described for the first time since by Gerald Oster , that include the presentation of two acoustic stimuli with similar frequencies through the two channels of stereo headphones. The interference of their waves which occurs at the level of the central nervous system, produces a composite signal with a frequency resulting from the difference of the two original frequencies. For example if you give an acoustic stimulus of 100 Hz to an ear and simultaneously administering another acoustic stimulation of 104 Hz to the opposite ,ear the person who listens to these stimuli will perceive a "Binaural Beat" of 4 Hz caused by the difference between the two frequencies.

These Binaural Beats are of interest because they have been thought to cause hemispheric synchronization and influence the EEG frequency like light stimulation .

Binaural Beats have already been used in humans undergoing outpatient surgery in urogynecological and have been shown to help increase patient comfort by reducing the state of anxiety and pain without interfering negatively with postoperative functional recovery . In this study the investigators evaluate the use of Binaural Beat in outpatients to undergo colonoscopy to reduce pain .

A total of 100 patients divided into two groups, 50 treatment and 50 control will be considered.

Both patient groups will be invited to wear headphones regardless of whether they have been randomized to Binaural Beats with white noise or white noise only to ensure blindness of participation The headphones will be worn ten minutes before and throughout the procedure. Pain will be measured by VAS scale and satisfaction by Likert scale after the procedure in both groups. Blood pressure and heart rate will be monitored before, during, and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for outpatient colonoscopy
* Valid consent expression to the study participation
* Good collaboration in activities provided by the study

Exclusion Criteria:

* Insufficient degree of collaboration
* Abnormal hearing
* Denial of informed consent to participate in the study
* Previous colon resection surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Pain perception evaluated with VAS | 5 minutes after completing the procedure (complete withdrawal of the colonoscope)
  Comparison between the two groups of pain perceived during the procedure by VAS scale. The Visual Analogue Scale (VAS) is a validated scale for measuring pain on 11 points, from 0 to 10, in which the patient indicates the maximum perceived pain.

SECONDARY OUTCOMES:
Comparison between the two groups of the level of satisfaction: Likert scale | 5 minutes after completing the procedure (complete withdrawal of the colonoscope)
  Comparison between the two groups of the level of satisfaction of the entire procedure measured with a Likert scale . Likert scale is a scale which is used to allow the individual to express how much they agree or disagree with a particular statement patient satisfaction rated as: not at all, very low, moderate satisfaction, complete satisfaction; (b) willingness to repeat the procedure in the future:
  not at all, very low, barely yes, yes;
Blood pressure assessment | 3 minutes before inserting the colonoscope (this was baseline), 5 minutes after colonoscope insertion and 3 minutes after completing the procedure (complete withdrawal of the colonoscope);
  Systolic and diastolic blood pressure evaluation measured in millimeters of Hg
Heart rate assessment | 3 minutes before inserting the colonoscope (this was baseline), 5 minutes after colonoscope insertion and 3 minutes after completing the procedure (complete withdrawal of the colonoscope);
  Heart rate evaluation measured in beats/min.
comparison on the number of subjects who could not complete the exam | at the end of the planned study in a year
  comparison on the number of subjects between the two groups who could not complete the exam due to intolerance
comparison on the use of drugs during the procedure | at the end of the planned study in a year
  comparison between the two groups on the use of atropine during the procedure to reduce vagal effects

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Tani, MD, Principal Investigator — USL AREA VASTA TOSCANA NORDOVEST
Locations (1):
- Santa Maria Maddalena Hospital, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa A, Montalbano LM, Orlando A, Ingoglia C, Linea C, Giunta M, Mancuso A, Mocciaro F, Bellingardo R, Tine F, D'Amico G. Music for colonoscopy: A single-blind randomized controlled trial. Dig Liver Dis. 2010 Dec;42(12):871-6. doi: 10.1016/j.dld.2010.03.016. Epub 2010 May 7. PMID 20452299
- [Background] Wang MC, Zhang LY, Zhang YL, Zhang YW, Xu XD, Zhang YC. Effect of music in endoscopy procedures: systematic review and meta-analysis of randomized controlled trials. Pain Med. 2014 Oct;15(10):1786-94. doi: 10.1111/pme.12514. Epub 2014 Aug 19. PMID 25139786
- [Background] Rudin D, Kiss A, Wetz RV, Sottile VM. Music in the endoscopy suite: a meta-analysis of randomized controlled studies. Endoscopy. 2007 Jun;39(6):507-10. doi: 10.1055/s-2007-966362. PMID 17554644
- [Background] Lembo T, Fitzgerald L, Matin K, Woo K, Mayer EA, Naliboff BD. Audio and visual stimulation reduces patient discomfort during screening flexible sigmoidoscopy. Am J Gastroenterol. 1998 Jul;93(7):1113-6. doi: 10.1111/j.1572-0241.1998.00339.x. PMID 9672340
- [Background] Garcia-Argibay M, Santed MA, Reales JM. Efficacy of binaural auditory beats in cognition, anxiety, and pain perception: a meta-analysis. Psychol Res. 2019 Mar;83(2):357-372. doi: 10.1007/s00426-018-1066-8. Epub 2018 Aug 2. PMID 30073406
- [Background] Tani A, Vagheggini G, Moretti F, Del Colombo V, Lehle J, Campana S, Labate A, Tomaiuolo F. Binaural Beats Reduce Postoperative Morphine Consumption in Older adults After Total Knee Replacement Surgery. Altern Ther Health Med. 2021 Mar;27(2):27-30. PMID 32412916